CLINICAL TRIAL: NCT04617132
Title: Online Mindfulness Groups for Families Affected by Postpartum Depression and Anxiety: Study Protocol
Brief Title: Online MBI for Families Affected by PPDA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: British Columbia Children's Hospital (Other)
Responsible Party: Principal Investigator, Katarina Tabi, Research Fellow, British Columbia Children's Hospital
Other Study IDs: H20-01884
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Postpartum Depression; Postpartum Anxiety
Keywords: Mindfulness
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Online Mindfulness Group: Families with PPDA receiving evidence-based MBCT/MBSR intervention
  Interventions: Behavioral: MBCT/MBSR

INTERVENTIONS:
Behavioral: MBCT/MBSR — This intervention teaches the practice of mindfulness - being aware of the present moment without judgement - to help reduce the emotional reactivity to thoughts and bodily sensations, which prevents downward spirals into depression, anxiety, or fear.

SUMMARY:
The aim of this study is to explore the feasibility of delivering clinical mindfulness groups for families affected with postpartum depression and anxiety (PPDA). Families with PPDA are a vulnerable population who already face challenges during the postpartum period, but now the Covid-19 era has brought extra challenges - lower availability of family members or support systems to help in person, older children at home as childcare facilities are closed, etc. Clinical mindfulness groups are now being run online to support this population, with the current barriers of having to stay at home. Through this study, we want to capture the challenges that both clinicians and participants might face using virtual platforms (e.g. technical difficulties), to see whether online delivery of clinical mindfulness groups is feasible.

DETAILED DESCRIPTION:
Postpartum depression and anxiety (PPDA) is a prevalent condition, affecting about every 1 in 5 families. This not only impacts the parent diagnosed with PPDA but also affects relationships with the rest of the family, ability to bond with her child, and can cause tension between the parents. Thus, it is important that steps are taken to effectively treat and support families affected by PPDA in a timely manner. On top of the struggles with a newborn baby, the Covid era has brought along some new challenges. One such challenge is that many healthcare providers and clinics have limited capacities or the care they provide may be limited due to lockdown and Covid-19. Another challenge is the decreased in-person support from family and other support systems, as well as having older children at home all the time due to childcare facilities being closed.

As it is important to offer this population some support, this study is being conducted to see if continuing the clinical groups and turning them onto a distant, online format would be possible, and if it would work for both clinicians and the postpartum population.

The aim of the study is to determine the feasibility of running online clinical mindfulness groups, particularly examining whether patients are able to access and continue with the online sessions. Feasibility will be assessed by frequency of technical difficulties faced by patients or clinicians and number of disruptions or episodes of parents leaving their screens (e.g. to calm their child), self-report items of how participants found attending online sessions and following the program, and attendance and drop-out rates. Secondary outcomes of this study include reasons for drop-outs, satisfaction and acceptability, couple interactions, and mental health outcomes.

The mindfulness groups will be rooted in the evidence-based 8-week programs, including Mindfulness-Based Stress Reduction (MBSR) and Mindfulness-Based Cognitive Therapy (MBCT), and adapted for this population needs. The mindfulness groups will run once a week, totalling 8 sessions over the course of 8 weeks. These groups will be run by trained clinicians and mindfulness facilitators and will be a part of the RMH clinical program.

ELIGIBILITY:
Inclusion Criteria:

* Are able to read and write in English.
* Are in a cohabiting relationship - woman with PPDA and partner living together.
* Woman with PPDA has been diagnosed with MDD and/or GAD as per the DSM-5 criteria, up to 12 months postpartum.

Exclusion Criteria:

* Are younger than 19 years old.
* Women with PPDA assessed to currently have a substance use disorder, psychotic disorder, or suicidality.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Invited from a tertiary mental health clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Weekly (Week 1-8)
  Assessed via participant attendance and clinician survey about technological difficulties

SECONDARY OUTCOMES:
Acceptance & Satisfaction | Week 8
  Self-report questionnaire completed by participants
Relationship & Interactions | Week 1, 4, 8, and Follow-up
  This is a newly developed self-report measure that explores couple interactions and relationship satisfaction
PHQ-9 | Week 1, 4, 8, and Follow-up
GAD-7 | Week 1, 4, 8, and Follow-up

OTHER OUTCOMES:
Demographics | Week 1
  Demographics questionnaire sent to participants

CONTACTS AND LOCATIONS:
Overall Officials: S. Evelyn Stewart, Principal Investigator — British Columbia Children's Hospital
Locations (1):
- Reproductive Mental Health Program, BC Children's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Tabi K, Bhullar M, Fantu L, Shulman B, Dueck R, Hippman C, Ryan D, Stewart SE. Feasibility of online mindfulness-based interventions for families affected with postpartum depression and anxiety: study protocol. BMJ Open. 2022 Sep 7;12(9):e051935. doi: 10.1136/bmjopen-2021-051935. PMID 36691183